CLINICAL TRIAL: NCT04464395
Title: Immunotherapy of COVID-19 With B-Cell Activating CPI-006 Monoclonal Antibody
Brief Title: Study of CPI-006 as Immunotherapy for Hospitalized COVID-19 Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-006-002
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
Keywords: SARS CoV-2; Coronavirus; Covid
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — CPI-006; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPI-006 Dose Escalation (Experimental): CPI-006 + Standard of Care
  Interventions: Drug: CPI-006
- Control Arm (Other): Standard of Care Only
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: CPI-006 — Participants will receive a single dose of CPI-006 at one of four dose levels (0.3 mg/kg, 1.0 mg/kg, 3.0 mg/kg, or 5.0 mg/kg) along with standard of care.
  Arms: CPI-006 Dose Escalation
Other: Standard of Care — Participants will receive standard of care treatment only.
  Arms: Control Arm

SUMMARY:
This Phase 1 single-dose, dose-escalation study is an open label trial evaluating the safety of CPI-006, a humanized monoclonal antibody targeting the CD73 cell-surface ectonucleotidase, as immunotherapy for stable hospitalized mild or moderately symptomatic COVID-19 patients with a parallel non-randomized Control Arm for treatment with standard of care only.

ELIGIBILITY:
Inclusion Criteria:

* Nasal swab test positive by reverse transcriptase PCR for SARS CoV-2 within past 7 days, and onset of COVID-19 symptoms no more than 10 days prior to the positive test
* Hospitalized and have stable mild to moderate symptoms of COVID-19
* Blood oxygen saturation of a minimum of 92% on either no oxygen or up to 5L/min supplemental oxygen
* Patients with cancer must be in remission or have stable, controlled disease and may be actively receiving drugs or biologics not deemed by the investigator to likely affect immune response.
* Women must not be of child bearing potential or agree to use contraceptive guidance for 6 weeks

Exclusion Criteria:

* Patients receiving previous invasive mechanical ventilation or non-invasive ventilation (CPAP, BiPAP) for COVID-19 illness
* Patients hospitalized >7 days prior to receiving study intervention
* Other diseases or conditions that are not controlled
* On drugs or biologics that are immunosuppressive, cytotoxic or immunomodulatory
* Patients with autoimmune disease must be controlled on non immunosuppressive or immune modifying agents
* Have received cytotoxic, immunosuppressive or immunomodulatory agents within past 3 months (other than for treatment of COVID-19).
* Patients receiving experimental therapies that are immunosuppressive
* Patients receiving non-immuno-suppressive experimental therapies within 7 days prior to receiving CPI-006
* Patients receiving convalescent plasma within 24 hours prior to receiving CPI-006
* Patients receiving experimental anti-SARS CoV-2 monoclonal antibodies within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events to Determine Single Dose of CPI-006 That is Safe in Patients with COVID-19 | Up to 30 days after dose of CPI-006.
  Incidence of adverse events (including serious adverse events and dose limiting toxicities).
Immunoglobulin Anti-SARS CoV-2 Levels | Baseline and Day 28.
  Measure changes in serum or plasma immunoglobulin anti-SARS CoV-2 levels.

SECONDARY OUTCOMES:
Negative Nasal Swab Polymerase Chain Reaction (PCR) SARS CoV-2 Viral Tests | Baseline to two consecutive negative nasal swab PCR SARS CoV-2 viral tests (separated by at least 48 hours).
  Time to two consecutive negative nasal swab PCR SARS CoV-2 viral tests.
Duration of symptoms | Up to 24 weeks after dose of CPI-006.
  Duration of COVID-19 related symptoms.
Time to discharge | Up to 24 weeks after dose of CPI-006.
  Time to discharge from hospital.
Rate of medical procedures | Up to 24 weeks after dose of CPI-006.
  Rate of medical procedures during hospitalization.
Difference in changes in serum/plasma immunoglobulin anti-SARS CoV-2 levels | Baseline and visits through Day 28.
  Difference between Active Arm and Control Arm patients in terms of changes in serum or plasma immunoglobulin anti-SARS CoV-2 levels.

CONTACTS AND LOCATIONS:
Overall Officials: S. Mahabhashyam, MD. MPH, Study Chair — Corvus Pharmaceuticals
Locations (3):
- United States (3):
  - El Centro Regional Medical Center, El Centro, California
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Temple University Hospital, Philadelphia, Pennsylvania